CLINICAL TRIAL: NCT06304298
Title: The Neutrophil-to-lymphocyte Ratio (NLR) and Platelet-to-lymphocyte Ratio (PLR) Levels Following IPACK Block in Knee Arthroplasty: a Randomized, Controlled Trial.
Brief Title: NLR and PLR Levels Following IPACK Block in Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10/2023
Record Dates: First submitted 2023-05-24; First posted 2024-03-12 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Knee Arthropathy; Knee Osteoarthritis; Knee Pain Chronic
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Sodium Chloride; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham blocks (Active Comparator): iPACK block with 20ml of 0.9% sodium chloride
  Interventions: Drug: 0.9% Sodium Chloride Injection
- iPACK block (Active Comparator): iPACK block with 20ml 0f 0.2% ropivacaine
  Interventions: Drug: Ropivacaine 0.2% Injectable Solution

INTERVENTIONS:
Drug: 0.9% Sodium Chloride Injection — After spinal anesthesia, the ultrasound-guided iPACK block will be performed with 20ml of 0.9% sodium chloride
  Other Names: Placebo
  Arms: Sham blocks
Drug: Ropivacaine 0.2% Injectable Solution — After spinal anesthesia, the ultrasound-guided iPACK block will be performed with 20ml of 0.2% ropivacine
  Other Names: iPACK block
  Arms: iPACK block

SUMMARY:
Effect of iPACK block on NLR and PLR following knee arthroplasty

DETAILED DESCRIPTION:
The NLR is a sensitive indicator of inflammation confirmed in numerous studies and has a predictive and prognostic value. NLR is a cheap, simple, fast-acting, readily available stress and inflammation parameter with high sensitivity and low specificity. Dynamic changes in the NLR precede the clinical state for several hours and may alert clinicians early about the ongoing pathological process. NLR is a new promising marker of cellular immune activation, an important indicator of stress and systemic inflammation. It opens a new dimension for clinical medicine to understand better the biology of inflammation, the linkage, and antagonism between innate and adaptive immunity, and its clinical consequences for health and disease.

NLR is affected not only by surgical trauma but also by the method of anesthesia. In recent years, the influence of regional anesthesiology on reducing the inflammatory response after surgical procedures has been emphasized. However, there have been very few studies evaluating the effect of various methods of anesthesia on the NLR.

This is the first study to investigate the effect of regional anesthesia on the NLR and PLR in patients undergoing knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA classification I-III
* Aged 20-90 years
* Who will be scheduled for hip arthroplasty under spinal anesthesia

Exclusion Criteria:

* Patients who have a history of bleeding diathesis
* Take anticoagulant therapy
* History of chronic pain before surgery
* Multiple trauma
* patients unable to assess their pain (dementia)
* patients operated under general anesthesia
* patients having an infection in region of the procedure
* patient who do not accept the procedure

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Neutrophil-to-lymphocyte ratio | 12 hours after surgery
  Neutrophil to lymphocyte ratio (NLR) is used as a marker of subclinical inflammation. It is calculated by dividing the number of neutrophils by number of lymphocytes, usually from peripheral blood sample, but sometimes also from cells that infiltrate tissue, such as tumor.

SECONDARY OUTCOMES:
PLR | 12 hours after surgery
  Platelet-to-lymphocyte ratio
PLR | 24 hours after surgery
  Platelet-to-lymphocyte ratio
PLR | 48 hours after surgery
  Platelet-to-lymphocyte ratio
NLR | 24 hours after surgery
  Neutrophile-to-lymphocyte ratio
NLR | 48 hours after surgery
  Neutrophile-to-lymphocyte ratio
first need of opiate | 48 hours after procedure
  Time after surgery when the patient needs opiate for the first time
Opioid Consumption | 48 hours after surgery
  Total opiate consumption after surgery
Pain score | 4 hours after surgery
  NRS (Numerical Rating Scale)
Pain score | 8 hours after surgery
  NRS (Numerical Rating Scale)
Pain score | 12 hours after surgery
  NRS (Numerical Rating Scale)
Pain score | 18 hours after surgery
  NRS (Numerical Rating Scale)
Pain score | 24 hours after surgery
  NRS (Numerical Rating Scale)
Pain score | 36 hours after surgery
  NRS (Numerical Rating Scale)
Pain score | 48 hours after surgery
  NRS (Numerical Rating Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Domagalska, Ph.D., Principal Investigator — Poznań University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poznań, Poland

IPD SHARING:
Plan to Share IPD: No